CLINICAL TRIAL: NCT00272844
Title: Treatment of the Cholesterol Defect in Smith-Lemli-Opitz Syndrome
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Boston Children's Hospital (Other)
Responsible Party: Principal Investigator, Mira Irons, Associate Chief, Division of Genetics, Boston Children's Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 03-11-189R
Record Dates: First submitted 2006-01-04; First posted 2006-01-09 (Estimated); Results first posted 2017-10-20 (Actual); Last update posted 2017-10-20 (Actual); Status verified 2017-09

CONDITIONS: Smith-Lemli-Opitz Syndrome
Keywords: cholesterol; Smith-Lemli-Opitz syndrome; mental retardation; sterols; congenital anomalies
MeSH Terms: conditions — Smith-Lemli-Opitz Syndrome; Intellectual Disability; Congenital Abnormalities

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Cholesterol supplementation (Experimental)
  Interventions: Drug: crystalline cholesterol oil-based suspension

INTERVENTIONS:
Drug: crystalline cholesterol oil-based suspension — 200 mg/mL suspension of crystalline cholesterol in oil. Dosage (generally 75-300 mg/kg/day in divided doses) is based on initial cholesterol levels and regulated to increase, yet maintain, cholesterol levels no higher than normal ranges.

SUMMARY:
The purpose of this study is to determine whether supplementation with an oil-based cholesterol suspension will correct the biochemical abnormalities in cholesterol and its precursors in individuals with the Smith-Lemli-Opitz syndrome.

DETAILED DESCRIPTION:
This study involves treating individuals with the Smith-Lemli-Opitz syndrome, a rare inborn error of cholesterol metabolism, with supplemental cholesterol to determine it effects on biochemical sterol metabolites, growth, neuropsychological development, ophthalmologic and auditory function, ERG (electroretinogram) parameters, and CNS metabolites as determined by brain MRS-imaging. Safety of the supplemental cholesterol suspension is monitored by tests of hematologic, renal, and liver function at periodic intervals. There is also a substudy that is investigating potential genotype-phenotype correlations, as well as another that studies biochemical parameters of light sensitivity in cultured skin fibroblasts from affected patients.

ELIGIBILITY:
Inclusion Criteria:

* Biochemical confirmation of sterol defect associated with Smith-Lemli-Opitz syndrome

Exclusion Criteria:

* Inability to tolerate crystalline cholesterol
* Inability to travel to Boston 3-4 times/year based on age

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 1998-01; Primary Completion 2011-06 (Actual); Study Completion 2011-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mira Irons, M.D., Principal Investigator — Boston Children's Hospital
Locations (1):
- Children's Hospital Boston, Boston, Massachusetts, United States

REFERENCES:
- [Result] Irons M, Elias ER, Tint GS, Salen G, Frieden R, Buie TM, Ampola M. Abnormal cholesterol metabolism in the Smith-Lemli-Opitz syndrome: report of clinical and biochemical findings in four patients and treatment in one patient. Am J Med Genet. 1994 May 1;50(4):347-52. doi: 10.1002/ajmg.1320500409. PMID 8209913
- [Result] Elias ER, Irons MB, Hurley AD, Tint GS, Salen G. Clinical effects of cholesterol supplementation in six patients with the Smith-Lemli-Opitz syndrome (SLOS). Am J Med Genet. 1997 Jan 31;68(3):305-10. doi: 10.1002/(sici)1096-8628(19970131)68:33.0.co;2-x. PMID 9024564
- [Result] Irons M, Elias ER, Abuelo D, Bull MJ, Greene CL, Johnson VP, Keppen L, Schanen C, Tint GS, Salen G. Treatment of Smith-Lemli-Opitz syndrome: results of a multicenter trial. Am J Med Genet. 1997 Jan 31;68(3):311-4. PMID 9024565
- [Result] Caruso PA, Poussaint TY, Tzika AA, Zurakowski D, Astrakas LG, Elias ER, Bay C, Irons MB. MRI and 1H MRS findings in Smith-Lemli-Opitz syndrome. Neuroradiology. 2004 Jan;46(1):3-14. doi: 10.1007/s00234-003-1110-1. Epub 2003 Nov 5. PMID 14605787
- [Result] Elias ER, Hansen RM, Irons M, Quinn NB, Fulton AB. Rod photoreceptor responses in children with Smith-Lemli-Opitz syndrome. Arch Ophthalmol. 2003 Dec;121(12):1738-43. doi: 10.1001/archopht.121.12.1738. PMID 14662594

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients newly diagnosed with Smith-Lemli-Opitz syndrome at Boston Children's Hospital were offered enrollment in the study from 1998 until it's completion. The study was completed and closed to enrollment here in June, 2010 and the IND was withdrawn in July, 2011.
Groups:
- Cholesterol Supplementation: crystalline cholesterol oil-based suspension : 200 mg/mL suspension of crystalline cholesterol in oil. Dosage (generally 75-300 mg/kg/day in divided doses) is based on initial cholesterol levels and regulated to increase, yet maintain, cholesterol levels no higher than normal ranges.
Period: Overall Study
Arm/Group | Cholesterol Supplementation
Started | 23
Completed | 18
Not Completed | 5
Not completed — Withdrawal by Subject | 5

BASELINE CHARACTERISTICS:
Population: All patients had elevation of 7-DHC diagnostic of SLOS
Arm/Group | Cholesterol Supplementation
Number analyzed (Participants) | 23
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 18
  Between 18 and 65 years | 5
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12
  Male | 11
Region of Enrollment [Number; unit: participants]
  United States | 23

OUTCOME MEASURES:

1. Primary Outcome: Number of Responders
Description: Responders was defined as an increase in total serum cholesterol and a decrease in 7-DHC (7-Dehydrocholesterol), and 8-DHC (8-Dehydrocholesterol) were measured on all participants.
Time Frame: Every 3-6 months for an approximate median of 5 years
Measure: Count of Participants; unit: Participants
Arm/Group | Cholesterol Supplementation
Number analyzed (Participants) | 18
Participants | 18

2. Secondary Outcome: Number of Growth Responders
Description: Growth response was defined as an increase in general health, growth, and behavior.
Time Frame: Every 3-6 months for an approximate median of 5 years
Measure: Count of Participants; unit: Participants
Arm/Group | Cholesterol Supplementation
Number analyzed (Participants) | 18
Participants | 18

3. Secondary Outcome: Number of Participants With Improved Neuropsychological Development
Description: Improved neuropsychological development is defined as progressively achieving developmental milestones
Time Frame: Every 3-6 months for an approximate median of 5 years
Measure: Count of Participants; unit: Participants
Arm/Group | Cholesterol Supplementation
Number analyzed (Participants) | 18
Participants | 18

ADVERSE EVENTS:
Arm/Group | Cholesterol Supplementation
Serious Adverse Events (participants affected / at risk) | 0/23
Other Adverse Events (participants affected / at risk) | 0/23

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes